CLINICAL TRIAL: NCT04336007
Title: Effects of Diathermy Application on Immediate Sports Performance of Paralympic Swimmers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20/135-E_TFM
Record Dates: First submitted 2020-03-24; First posted 2020-04-07 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2020-03

CONDITIONS: Athletic Performance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Radio-frequency group (Experimental): The equipment used, INDIBA® Activ Ct9, (448kHz), with the switch-mode on.
  Interventions: Device: Resistive Diathermy (INDIBA® Activ Ct9)
- Placebo group (Placebo Comparator): The equipment used, INDIBA® Activ Ct9, (448kHz), with the switch-mode off.
  Interventions: Device: Resistive Diathermy OFF (INDIBA® Activ Ct9)
- Control Group (Sham Comparator): NO INTERVENTION athlete's usual pre-competition warming-up
  Interventions: Other: Control

INTERVENTIONS:
Device: Resistive Diathermy (INDIBA® Activ Ct9) — Intervention is conducted using a 65-mm diameter Resistive (RES) electrode (movable), and a planar electrode was used as a return electrode on the abdomen. The electricity is administered in the following manner: cream was applied to the upper limbs existent area, and the electrical output is marked at 75% by moving the movable electrode and if not tolerated by the patient lowered until 35%, Therapy is conducted for 20 minutes, prior swimming time trials.
  Arms: Radio-frequency group
Device: Resistive Diathermy OFF (INDIBA® Activ Ct9) — Placebo is conducted using a 65-mm diameter RES electrode (movable), and a planar electrode was used as a return electrode on the abdomen. The electricity IS NOT administered, the cream was applied to the upper limbs existent area and moving the movable electrode, intervention is conducted for 20 minutes, prior to swimming time trials.
  Arms: Placebo group
Other: Control — This group will warm-up as they usually do in competitions, for later time trial measuring.
  Arms: Control Group

SUMMARY:
This study aims to evaluate the potential benefits of Monopolar Capacitive Resistive Radio-frequency (448 kHz) on the sports performance of Paralympic swimmers.

DETAILED DESCRIPTION:
A randomized, double-blind, crossover, controlled and sham-controlled clinical trial

Evaluate the effectiveness of resistive capacitive diathermy as sports performance enhancement of Paralympic elite swimmers compared with a "sham" diathermy treatment and with a control group. The resistive capacitive diathermy is a medical device supplying low (448 kHz) radiofrequency with a maximum output power of 200 W, used to improve physiological aspects and theoretically allowing improvement in swimming performance. The sham diathermy treatment is administered with the device set on "on" but not active (not supplying energy) and control group will not receive anything, randomly assigned to either resistive capacitive diathermy treatment (group 1), sham-treatment (group 2) or control (group 3) athletes are submitted to a twenty minutes session prior swimming performance. The main outcome measures are the simulate swimming time trial (seconds) to assess time completing the presented course and Borg Scale for perceived exertion. Outcome measures are administered at completing each time trial.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent signed.
* Age between 18 y 70 years old.
* Already in the position of the International Paralympic Committee (IPC) classification.
* Know their personal mark (50-100mts).
* Having the capacity to fill and understand questionnaires, understand and follow verbal orders.

Exclusion Criteria:

* Pregnancy.
* Use of pacemakers or other types of electronic implants
* Non-intact skin (open wounds or recent burns)
* thrombophlebitis
* Known allergy to nickel and chromium
* Symptomatic anemia (hemoglobin below 12g / dl presenting any of these symptoms: tiredness, shortness of breath, dizziness, palpitations or headache).
* Present feverish process

Elimination criteria:

* Revocation of inform consent.
* Attend to less than three visits.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2020-03-16 (Actual); Primary Completion 2021-05 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Time-trials (Experimental Group) | through study completion, an average of 4 months
  Time in Seconds that takes the athlete since taking off from the edge of the pool until reaching two different distances, 50 and 100 meters, measuring each distance twice, time will be measure by technical digital chronometer.
Time-trials (Placebo Group) | through study completion, an average of 4 months
  Time in Seconds that takes the athlete since taking off from the edge of the pool until reaching two different distances, 50 and 100 meters, measuring each distance twice, time will be measure by technical digital chronometer.
Time-trials (Sham Group) | through study completion, an average of 4 months
  Time in Seconds that takes the athlete since taking off from the edge of the pool until reaching two different distances, 50 and 100 meters, measuring each distance twice, time will be measure by technical digital chronometer.
Change of Perceived exertion (Experimental Group) | through study completion, an average of 4 months
  To measure the athlete's qualification of their exertion the Borg Rate of Perceived Exertion (RPE) Scale® will be used, previously validated and with the proper license, measures will be taken pre/post-competition.
Change of Perceived exertion (Placebo group) | through study completion, an average of 4 months
  To measure the athlete's qualification of their exertion the Borg Rate of Perceived Exertion (RPE) Scale® will be used, previously validated and with the proper license, measures will be taken pre/post-competition.
Change of Perceived exertion (Sham group) | through study completion, an average of 4 months
  To measure the athlete's qualification of their exertion the Borg Rate of Perceived Exertion (RPE) Scale® will be used, previously validated and with the proper license, measures will be taken pre/post-competition.

SECONDARY OUTCOMES:
Age | through study completion, an average of 4 months
  Birth date collected from the questionaire
Sex | through study completion, an average of 4 months
  Man or Woman
International Paralympic Committee Classification. | through study completion, an average of 4 months
  Code between S1-10, S11-13 or S14
Weight. | through study completion, an average of 4 months
  Weight in kilograms
Height. | through study completion, an average of 4 months
  Height in centimeters
Daily training time. | through study completion, an average of 4 months
  Time of training comprehended on the following intervals 0-3 hours/3-6 hours/>6hours
Comorbidity | through study completion, an average of 4 months
  Presence of different conditions that might interfere with the study.
Best swimming stroke | through study completion, an average of 4 months
  Choose between breaststroke, butterfly stroke, front crawl or backstroke.
Personal mark 50 mts. | through study completion, an average of 4 months
  Best time record for 50 meters distance
Personal mark 100 mts. | through study completion, an average of 4 months
  Best time record for 100 meters distance

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Garcia Fernández, Study Chair — Universidad Complutense de Madrid
Locations (1):
- Universidad Complutense de Madrid, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Sousa-De Sousa L, Espinosa HG, Mate-Munoz JL, Lozano-Estevan MDC, Cerrolaza-Tudanca S, Rozalen-Bustin M, Fernandez-Carnero S, Garcia-Fernandez P. Effects of Capacitive-Resistive Electric Transfer on Sports Performance in Paralympic Swimmers: A Stopped Randomized Clinical Trial. Int J Environ Res Public Health. 2022 Nov 7;19(21):14620. doi: 10.3390/ijerph192114620. PMID 36361500